CLINICAL TRIAL: NCT00784355
Title: Does Laparoscopic Cholecystectomy Prevent Recurrence in Idiopathic Pancreatitis? A Prospective Multicentre Randomized Study
Brief Title: Laparoscopic Cholecystectomy in Idiopathic Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Hannu Paajanen, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5200616
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Pancreatitis
Keywords: recurrence of idiopathic pancreatitis; laparoscopic cholecystectomy; etiology of pancreatitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic; Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:Laparoscopic cholecystectomy (Experimental): Surgery
  Interventions: Procedure: Laparoscopic cholecystectomy
- 2:controls (No Intervention): non-surgical control group

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Surgery
  Other Names: idiopathic pancreatitis; cholecystectomy
  Arms: 1:Laparoscopic cholecystectomy

SUMMARY:
The causes of acute pancreatitis in Finland are alcohol overuse (60%), cholecystolithiasis (20%) and idiopathic (i.e. etiology unknown)(20%). Acute pancreatitis may recur in over half of cases and may be fatal in severe cases in 30%. Majority of idiopathic pancreatitis are caused by microlithiasis in gall bladder. The purpose of this randomized study is to prevent recurrence of idiopathic pancreatitis by performing laparoscopic cholecystectomy compared to non-operative group in 2 years follow-up of patients.

DETAILED DESCRIPTION:
Etiologic investigations include serum amylase, lipase, triglyceride and calcium determination, as well as abdominal ultrasound scanning. Alcohol consumption is asked by using WHO audit test. After etiology of acute pancreatitis has been confirmed as idiopathic, 100 patients are randomized to laparoscopic cholecystectomy and 100 patients to follow-up of 2 years. Five to seven Finnish university and main central hospitals are participating the study.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic pancreatitis

Exclusion Criteria:

* age < 18 years old
* patients' refusal
* high operative risks
* alcohol overuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
recurrence of acute pancreatitis | 2 years

SECONDARY OUTCOMES:
etiology of acute pancreatitis in Finland in 2009-10 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karne S, Gorelick FS. Etiopathogenesis of acute pancreatitis. Surg Clin North Am. 1999 Aug;79(4):699-710. doi: 10.1016/s0039-6109(05)70036-0. PMID 10470320
- [Derived] Raty S, Pulkkinen J, Nordback I, Sand J, Victorzon M, Gronroos J, Helminen H, Kuusanmaki P, Nordstrom P, Paajanen H. Can Laparoscopic Cholecystectomy Prevent Recurrent Idiopathic Acute Pancreatitis?: A Prospective Randomized Multicenter Trial. Ann Surg. 2015 Nov;262(5):736-41. doi: 10.1097/SLA.0000000000001469. PMID 26583660